CLINICAL TRIAL: NCT00213642
Title: Value of Tc-99m Renography for Early Diagnosis of Cisplatin-induced Renal Toxicity
Brief Title: Tc-99m Renography and Cisplatin-induced Nephrotoxicity
Status: Terminated | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2000/003/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Cancer; Drug Toxicity; Kidney Failure
Keywords: Technetium Tc 99m Mertiatide; Radionuclide Imaging; Cisplatin; Kidney failure; Drug Toxicity; Cancer
MeSH Terms: conditions — Neoplasms; Drug-Related Side Effects and Adverse Reactions; Renal Insufficiency

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cisplatin is a heavy-metal complex widely used in the treatment of a variety of malignancies, including small cell and non-small cell lung cancer, ovarian, bladder, head and neck, esophageal, cervical and germ cell tumors. The administration of cisplatin is commonly associated with certain drug-induced toxicities that may limit their clinical utility and adversely affect the quality of life of patients undergoing treatment. Although many advances have been made in reducing some of the toxicities associated with platinum drug therapy, it is clear that dose-limiting nephrotoxicity remains a major stumbling block in the use of this compound. Subtle changes in renal function occur without overt renal insufficiency, consisting of a decrease in effective renal plasma flow and tubular dysfunction despite aggressive hydratation. Early tubular damage occurring within 1 to 3 hours after cisplatin administration has been demonstrated by measurement of urinary beta 2-microglobulin, a sensitive marker of tubular injury. The chronic lesion has become of greater concern in recent years as many patients have been cured or placed into long-term remission due to cisplatin treatment. It consists of a decrease in glomerular filtration rate, which is not necessary characterized by a remarkable increase in serum creatinine. Cumulative tubular damage has been demonstrated by increased urinary excretion of tubular enzymes such as alanine aminopeptidase and beta 2-microglobulin. In this setting, predicting the occurrence of chronic cisplatin-induced nephrotoxicity remains a clinical challenge.

Tc-99m mercaptoacetyltriglycine (MAG3) is predominantly a proximal tubular secretion renal agent without cortical fixation indicated for dynamic renal studies to evaluate cortical tubular function and collecting system drainage. Tc-99m MAG3 and is the agent of choice for obstructive uropathy and diffuse functional abnormalities of the renal cortex. The aim of this study was to evaluate by means of Tc-99m MAG3 scintigraphy the acute and subacute impairment of tubular secretion after cisplatin administration in patients with head and neck cancer receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck cancer
* Receiving a chemotherapy including cisplatin administration (>80 mg/m2)
* WHO score < or = 2
* Estimated life expectancy > 6 month
* Normal renal function
* Signed informed consent

Exclusion Criteria:

* Congestive heart failure
* History of cisplatin treatment
* Metastatic carcinoma
* History of radiation therapy
* History of renal insufficiency
* History of chronic renal disease
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-07; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Alain Manrique, MD, Study Chair — University Hospital, Rouen